CLINICAL TRIAL: NCT03563521
Title: Serum Cytokine Profiles of Severe Asthma
Brief Title: Identifying Serum Cytokine Profiles of Distinct Inflammatory Phenotypes in Severe Asthma
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Murat Türk, Principal Investigator, TC Erciyes University
Other Study IDs: astimsitokin
Record Dates: First submitted 2018-06-09; First posted 2018-06-20 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Asthma Persistent; Asthma, Allergic; Eosinophilic Asthma; Chronic Rhinosinusitis (Diagnosis)
Keywords: severe asthma; inflammatory phenotypes; serum cytokines; eosinophilia; atopy; chronic rhinosinusitis with nasal polyposis
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia; Disease; Eosinophilia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Serum nasopharyngeal brush (to detect pharyngeal tract pathogens with PCR)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Atopic, eosinophilic
- Atopic, non-eosinophilic
- Non-atopic, eosinophilic
- Chronic rhinosinusitis with/without nasal polyposis
- Non-atopic, non-eosinophilic
- Control: Without asthma, atopy and eosinophilia

SUMMARY:
The aim of this study is to determine and compare serum cytokine levels of six different severe asthma inflammatory phenotypes differentiated by their atopy, peripheral eosinophilia and/or chronic rhinosinusitis and/or nasal polyposis status.

DETAILED DESCRIPTION:
A prospective observational study of 90 adults diagnosed with severe asthma and on regular follow-up and 15 control subjects will be investigated. Stable (controlled or partly-controlled) status (of all) and exacerbated-status (if any) serum cytokine levels [IL-4, IL-5, IL-10, IL-13, IL-25, IL-33, thymic stromal lymphopoietin (TSLP), IL-17A, periostin) will be evaluated. Also nasopharyngeal brush samples will be obtained for respiratory tract panel work-up with PCR in exacerbated patients. Effect of viral infections' on cytokine response in different inflammatory phenotypes will be evaluated.

ELIGIBILITY:
Inclusion Criteria (for disease groups):

1. Patients diagnosed with severe asthma and followed-up at least 6 months at our clinic
2. Asthma that can only be complete or partly controlled with Global Initiative for Asthma (GINA) 4-5 treatment
3. Asthmatics that are eligible for the defined phenotypes
4. At least one perennial allergen sensitivity for the atopic groups

Inclusion Criteria (for control group):

1. Non-asthmatics (without clinical and pulmonary function test evidence)
2. Non-atopics (proved by skin prick tests)
3. Serum eosinophil count <300/cells

Exclusion Criteria (for disease groups):

1. <18 year-old
2. Smoking history within the last 1 year prior to the study
3. Asthmatics with inadequate inhaler technique and/or adherence problems
4. Comorbidities: malignancy history, connective tissue disorders, rheumatological disorders, hyperthyroidism, coronary heart diseases, diabetes mellitus, active hepatic diseases, akut kidney injury, any autoimmune diseases
5. Organ transplantation history
6. Pregnancy
7. Other pulmonary problems: chronic obstructive pulmonary disease (COPD), bronchiectasis, interstitial lung diseases, pulmonary thromboemboli
8. During stable period investigation

   1. Asthma control test <20
   2. Upper respiratory tract infections within 1 month before admission
   3. Exacerbation and/or systemic steroid use within 1 month before admission
9. Atopic patients that only have seasonal allergen sensitivity

Inclusion Criteria (for control group):

1. <18 year-old
2. Smoking history within the last 1 year prior to the study
3. Asthmatics with inadequate inhaler technique and/or adherence problems
4. Comorbidities: malignancy history, connective tissue disorders, rheumatological disorders, hyperthyroidism, coronary heart diseases, diabetes mellitus, active hepatic diseases, akut kidney injury, any autoimmune diseases
5. Organ transplantation history
6. Pregnancy
7. Other pulmonary problems: COPD, bronchiectasis, interstitial lung diseases, pulmonary thromboemboli
8. Without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asthmatic groups will be selected from the Erciyes University Allergy Clinic admisisons.
  Control group wil be selected from the Erciyes University Allergy Clinic admisisons and from the volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Serum cytokine levels | 10 months
  Measurement of stable state and exacerbation state levels of serum cytokines (IL-4, IL-5, IL10, IL-13, IL-17, IL-25, IL-33, TSLP, periostin)

SECONDARY OUTCOMES:
Nasal brush sample PCR | 10 months
  Detecting pharyngeal pathogens with PCR taken during exacerbated state

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University School of Medicine Division of Allergy, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided